CLINICAL TRIAL: NCT05901935
Title: A Multicentre, Randomized, Open-label, Controlled Phase Ш Clinical Study to Evaluate the Efficacy and Safety of DP303cversus Trastuzumab Combined With Vinorelbine/Capecitabine in of HER2-positive Advanced Breast Cancer
Brief Title: DP303c in Patients With HER2-positive Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1501-007
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: HER2-positive Advanced Breast Cancer
MeSH Terms: interventions — Trastuzumab; Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DP303c (Experimental): Eligible patients will be treated with DP303c at 3.0 mg/kg every 3 weeks.
  Interventions: Drug: DP303c
- Trastuzumab combined with vinorelbine/capecitabine (Active Comparator): Eligible patients will be treated with trastuzumab IV on day 1 and oral capecitabine twice daily on days 1-14 every 3 weeks, or patients will be treated with trastuzumab IV on day 1 and vinorelbine IV over on days 1 and 8 every 3 weeks.
  Interventions: Drug: Trastuzumab; Drug: Vinorelbine Tartrate; Drug: Capecitabine tablets

INTERVENTIONS:
Drug: DP303c — DP303c injection, 3.0 mg/kg, Q3W.
  Arms: DP303c
Drug: Trastuzumab — IV, 6 mg/kg, D1, Q3W
  Arms: Trastuzumab combined with vinorelbine/capecitabine
Drug: Vinorelbine Tartrate — IV, 25 mg/m^2，D1、D8，Q3W
  Arms: Trastuzumab combined with vinorelbine/capecitabine
Drug: Capecitabine tablets — PO 1000 mg/m^2, bid, D1-D14, Q3W
  Arms: Trastuzumab combined with vinorelbine/capecitabine

SUMMARY:
This is a study of DP303c in patients with HER2-positive advanced breast cancer.

DETAILED DESCRIPTION:
This is a multi-centre, randomized, open-label, controlled phase Ш clinical study to evaluate the efficacy and safety of DP303c injection versus trastuzumab combined with vinorelbine/capecitabine in the treatment of HER2-positive advanced breast cancer. Patients will be treated with DP303c injection at 3.0 mg/kg or trastuzumab combined with vinorelbine/capecitabine every 3 weeks. Patients will continue to receive treatment until disease progression, intolerable toxicity, withdrawal of informed consent, death, or any other reasons for treatment discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign the informed consent;
2. Age≥18 years old;
3. Patients with unresectable locally advanced or metastatic breast cancer confirmed by histology or cytology;
4. Confirmed to be HER2 positive by central lab (HER2-positive is defined as IHC 3+ or IHC 2+ with ISH positive);
5. Received at least 2 lines of systemic therapy for unresectable locally advanced, recurrent, or metastatic diseases;
6. Radiographic evidence of disease progression confirmed by the investigator during or after the most recent systemic treatment;
7. At least one assessable lesion at the baseline;
8. The Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
9. Patients with adequate organ function;
10. Life expectancy ≥ 12 weeks;
11. Female and male patient of childbearing age must agree to take adequate contraceptive measures during the entire study period.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. History of any other malignant tumors within three years
3. Has not recovered from adverse reactions caused by previous anti-tumor treatments to ≤ grade 1 or baseline (refer to NCI CTCAE 5.0);
4. The presence of active inflammatory bowel disease, chronic diarrhoea, short bowel syndrome or history of other gastrointestinal diseases or treatments that may affect intestinal absorption;
5. Received systemic anti-tumor therapy within 28 days before randomization, traditional Chinese medicine treatment with tumor indications approved by the National Medical Administration (NMPA) and palliative radiotherapy within 2 weeks before randomization;
6. Major organ surgery (excluding needle biopsy) within 28 days before randomization;
7. The cumulative amount of previous exposure to anthracyclines has reached the dosage;
8. Untreated (including baseline findings) or unstable cerebral parenchymal metastasis, spinal cord metastasis or compression, and cancerous meningitis.
9. History of LVEF < 40%, symptomatic congestive heart failure (CHF),.
10. Serious or uncontrolled cardiovascular disease;
11. History of (non-infectious) interstitial lung disease/pneumonitis requiring steroid hormone therapy;
12. Patients who currently have corneal diseases that require medication or surgical intervention;
13. Peripheral neuropathy ≥ grade 3 (refer to NCI CTCAE 5.0);
14. Active infections requiring intravenous antibiotics, antivirals, or antifungals within 2 weeks before randomization;
15. Active hepatitis B or C;
16. History of immunodeficiency diseases, including human immunodeficiency virus (HIV) positive;
17. Known hypersensitivity or contraindication to the active ingredients or excipients of the study drugs;
18. Treated with strong CYP3A inhibitors or strong CYP3A inducers before randomization;
19. There are other circumstances that may interfere with the subject's participation in the study procedures or do not meet the subject's maximum benefit from participating in the study or affect the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by BIRC | Up to approximately 5 years
  PFS is evaluated by a Blinded Independent Review Committee (BIRC) according to the Response Evaluation Criteria for Solid Tumors (RECIST) V1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator | Up to approximately 5 years
  PFS is evaluated by investigator according to the Response Evaluation Criteria for Solid Tumors (RECIST) V1.1.
Overall Survival (OS) | Up to approximately 5 years
  Overall Survival
Objective response rate (ORR) | Up to approximately 5 years
  ORR is evaluated by investigator and BIRC according to the Response Evaluation Criteria for Solid Tumors (RECIST) V1.1.
Duration of response (DoR) | Up to approximately 5 years
  Duration of Response
Incidence and severity of adverse events (AEs) | Up to approximately 5 years
  Incidence and severity of adverse events

IPD SHARING:
Plan to Share IPD: No